CLINICAL TRIAL: NCT02310425
Title: A Single Blinded Study on the Effect of Saccharomyces Boulardii CNCM I-745 on Growth and Development in Preterm Infants
Acronym: SBP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lingfen Xu, MD (Other)
Responsible Party: Sponsor-Investigator, Lingfen Xu, MD, A single blinded study on the effect of Saccharomyces boulardii CNCM I-745 on growth and development in preterm infants, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMU1
Record Dates: First submitted 2014-11-27; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases | interventions — Probiotics; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The study group (Active Comparator): The study group received S. boulardii supplementation, 50 mg/kg twice daily, compared to no intervention in the control group.
  Interventions: Drug: S. boulardii
- The control group (Placebo Comparator): A prospective, Placebo Comparator,randomized case-controlled trial was conducted in infants with a gestational age of 30 to 37 weeks and a birth weight between 1500 to 2500 g.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S. boulardii — 50 mg/kg twice daily
  Other Names: probiotics
  Arms: The study group
Drug: Placebo — he control group (group C) did not receive S. boulardii (nor other probiotics)
  Other Names: control group
  Arms: The control group

SUMMARY:
Immature gastrointestinal functions increase the risk of poor growth as well as nosocomial infections and necrotizing enterocolitis (NEC) in the preterm infant. The effects of probiotics on growth and development in premature infants have been investigated poorly. Saccharomyces boulardii CNCM I-745 (S. boulardii) is a non-pathogenic probiotic yeast.

Prophylactic supplementation of S. boulardii at a dose of 50 mg/kg twice a day appeared to bring preterm infants weight gain closer to that of intra-uterine growth rate, reduce feeding intolerance, and had no adverse effects.

DETAILED DESCRIPTION:
The objective of this study is to evaluate if feeding supplemented with S. boulardii can improve growth and clinical outcomes in preterm and low birth weight infants.

A prospective, randomized case-controlled trial was conducted in infants with a gestational age of 30 to 37 weeks and a birth weight between 1500 to 2500 g. The study group received S. boulardii supplementation, 50 mg/kg twice daily, compared to no intervention in the control group. The primary outcomes were short term growth parameters including weight gain, linear growth, head and chest circumference, and secondary outcomes were clinical outcomes, feeding intolerance and complications.

A total of 125 infants were enrolled in the study, 63 in the treatment and 62 in the control group. S. boulardii was administered for the first time at 2.63 days after birth (1 day to 6 days, 46 within 3 days, only 5 between 4 and 6 days).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were hospital born infants with a gestational age of 30 to 37 weeks and a birth weight between 1500 to 2500 g.

Exclusion Criteria:

* Exclusion criteria were severe neonatal pathology such as birth complications, GI malformations, chromosomal abnormalities, known immunodeficiency, hydrops foetalis, a central venous catheter and the use of antifungal drugs or probiotics.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
weight | The study period ended at the 28th day after birth or when the infant was discharged from the hospital if earlier, but the total period of the study was at least 7 days.
  weight gain (g/d)

SECONDARY OUTCOMES:
days of parenteral nutrition to full enteral nutrition | The study period ended at the 28th day after birth or when the infant was discharged from the hospital if earlier, but the total period of the study was at least 7 days.
  count the days of parenteral nutrition to full enteral nutrition
maximal enteral feed | The study period ended at the 28th day after birth or when the infant was discharged from the hospital if earlier, but the total period of the study was at least 7 days.
  measure maximal enteral feed (ml/day)
fasting time | The study period ended at the 28th day after birth or when the infant was discharged from the hospital if earlier, but the total period of the study was at least 7 days.
  count fasting time (days)
duration of hospitalisation | The study period ended at the 28th day after birth or when the infant was discharged from the hospital if earlier, but the total period of the study was at least 7 days.
  count the duration of hospitalisation (days)

OTHER OUTCOMES:
linear | The study period ended at the 28th day after birth or when the infant was discharged from the hospital if earlier, but the total period of the study was at least 7 days.
  linear growth (cm/week)
head circumference | The study period ended at the 28th day after birth or when the infant was discharged from the hospital if earlier, but the total period of the study was at least 7 days.
  head circumference growth (cm/week)
chest circumference | The study period ended at the 28th day after birth or when the infant was discharged from the hospital if earlier, but the total period of the study was at least 7 days.
  chest circumference growth (cm/week).